CLINICAL TRIAL: NCT05840146
Title: Effects of Kinesiotaping in Patients With Legg-Calvé-Perthes Disease: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Kineesiotaping for Patients With LCPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sezen Karaborklu Argut, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20151704-1746
Record Dates: First submitted 2023-03-20; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Legg-Calve-Perthes Disease
Keywords: Kinesiotape; Taping; Pediatric pain; Hip joint; Physiotherapy
MeSH Terms: conditions — Legg-Calve-Perthes Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotaping group (Experimental): Kinesiotape was applied to the lateral side of the affected hip for gluteus medius muscle. Each patient was positioned lying down with the affected side up, and two I-strips were used.
  Interventions: Other: Kinesiotaping
- Sham taping group (Sham Comparator): Sham tape was applied with a single I-strip without tension in tape or muscle stretch. After paper backing was completely removed, tape was essentially placed on the skin across the lateral side of the affected hip.
  Interventions: Other: Sham taping

INTERVENTIONS:
Other: Kinesiotaping — Two I-strips were used:
  1. The first-third of one I-strip began at the posterior iliac crest, without tension as an anchor. Then the patient actively flexed and adducted the affected hip, thus, the middle-third of the tape was applied with approximately 50% tension. Then the hip was set in its original position and the last-third of the tape ended approximately greater trochanter without tension.
  2. The first-third of the second I-strip was applied starting at the anterior iliac crest, without tension as an anchor. The patient actively extended and adducted the affected hip, thus, the middle-third of the tape was applied with approximately 50% tension. Then the hip was set in its original position and the last-third of the tape ended approximately greater trochanter without tension.
  Arms: Kinesiotaping group
Other: Sham taping — A single I-strip without tension in tape or muscle stretch. After paper backing was completely removed, tape was essentially placed on the skin across the lateral side of the hip.
  Arms: Sham taping group

SUMMARY:
Kinesiotaping is increasingly being used as a complement to musculoskeletal pain management. This study aimed to evaluate the immediate clinical efficacy of kinesiotaping on pain and pain-related symptoms of Legg-Calvé-Perthes Disease (LCPD).

DETAILED DESCRIPTION:
Kinesio taping is increasingly being used as a complement to musculoskeletal pain management. A randomized, double-blind, placebo-controlled clinical trial was conducted. Activity-related hip pain, passive and pain limited hip range of motion, gluteus medius muscle strength, function and balance were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Having received unilateral LCPD diagnosis,
* Anterior hip pain minimum three points on 10-cm Visual Analog Scale (VAS) over the previous week,
* Having the following symptoms; weakness of gluteus medius muscle and patient-reported complaints on function or balance

Exclusion Criteria:

* Having a history of any other hip pathologies,
* Having allergy to polyacrylate adhesive,
* Having used analgesic medication within the previous three days.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Immediate Clinical Efficacy on Activity Related Hip | The change between T1 (baseline) to T2 (thirty minutes later from the application)
  Horizontal 10 cm VAS (0, no pain; 10, the worst pain ever possible)

SECONDARY OUTCOMES:
Immediate Clinical Efficacy on Hip Abduction ROM | The change between T1 (baseline) to T2 (thirty minutes later from the application)
  goniometric range of motion (ROM)
Immediate Clinical Efficacy on Functional Task Durations | The change between T1 (baseline) to T2 (thirty minutes later from the application)
  10-meters walk task duration (sec) and 10-step climbing task duration (sec)
Immediate Clinical Efficacy on Balance test durations | The change between T1 (baseline) to T2 (thirty minutes later from the application)
  One leg stance test duration (sec) and Tandem walk test duration (sec)
Immediate Clinical Efficacy on Gluteus medius muscle strength | The change between T1 (baseline) to T2 (thirty minutes later from the application)
  muscle strength by handheld dynamometer (Ibs)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)